CLINICAL TRIAL: NCT03749824
Title: Investigation of Psychophysiological Response to Aversive Stimuli Over Time With Omega-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale-NUS College (Other)
Responsible Party: Principal Investigator, Jean Liu, Assistant Professor, Yale-NUS College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: YNC-SASSI-Quanti-2
Record Dates: First submitted 2018-10-29; First posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Conduct Disorder; ADHD; Oppositional Defiant Disorder
MeSH Terms: conditions — Conduct Disorder; Attention Deficit Disorder with Hyperactivity; Oppositional Defiant Disorder | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega-3 (Experimental): Children in this group will be given 400 mg of DHA and 600 mg of EPA. Caregivers will be instructed to give two 500mg Omega-3 capsules twice a day, at breakfast and at the evening meal for 6 months. Parents will be seen by the attending on a monthly basis for standard treatment procedure.
  Interventions: Dietary Supplement: Omega-3
- Placebo Capsules (Placebo Comparator): Children in this group will be given two placebo capsules twice daily; at breakfast and at the evening meal for a total period of 6 months.
  Interventions: Dietary Supplement: Placebo Capsules

INTERVENTIONS:
Dietary Supplement: Omega-3 — Omega-3 supplement is a highly concentrated fish oil brain booster supplement that helps compensate for the neurocognitive and brain dysfunction which acts as a predisposition to antisocial and violent behaviour. Individuals with antisocial personality disorder have been found to show an 11% reduction in gray matter in the prefrontal cortex (Raine et al. 2001), and structural prefrontal impairments are hypothesised to result in disinhibition of limbic subcortical structures that give rise to aggressive behaviour. Omega-3 (specifically DHA) is known to play a key role in neuronal structure and function.
  Arms: Omega-3
Dietary Supplement: Placebo Capsules — Children in this group will be given two placebo capsules twice daily; at breakfast and at the evening meal for a total period of 6 months.
  Arms: Placebo Capsules

SUMMARY:
This study investigates the psychophysiological responses to aversive stimuli in a population of 133 children clinically diagnosed with conduct disorder (CD) and/or attention-deficit/hyperactivity disorder (ADHD). Participants were administered with either omega-3 or placebo for a period of 6 months and were exposed to three stimuli every three months: 1) a loud sound, 2) threatening photographs from the International Affective Picture System (IAPS), and 3) the Trier Social Stress Task (TSST). Participants' psychophysiological features of heart rate and galvanic skin conductance were measured and analyzed in relation to their omega-3/placebo condition clinical diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between ages 7 and 16 years
2. Subjects who fulfil all criteria for a DSM-IV diagnosis of ADHD, conduct disorder, or oppositional defiant disorder
3. Subjects with willingness to participate in a randomized, double-blind controlled trial
4. Subjects with complete written, informed parental consent and child assent
5. Subjects with IQ of 70 or more

Exclusion Criteria:

1. Subjects who have IQ in the below 70
2. Subjects who are younger than 7 years old or older than 16 years old
3. Those without written parental consent
4. Those with brain pathology such as serious head injury, epilepsy, etc.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 133 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Heart Rate at 6 months | 7 minutes each at 0 months and 6 months
  For Trier Social Stress Task
Change from Baseline Skin Conductance Response at 6 months | 4 minutes each at 0 months and 6 months
  For loud sound
Change from Baseline Skin Conductance Response at 6 months | 4 minutes each at 0 months and 6 months
  For threatening photographs

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fung, Study Director — Institute of Mental Health, Singapore

IPD SHARING:
Plan to Share IPD: No